CLINICAL TRIAL: NCT07398378
Title: Clinical Investigation of Oral Malodor for Max Fresh Toothpaste Containing Zinc Citrate Versus a Commercially Available Regular Fluoride Toothpaste Using the Organoleptic Method: a Three-week Study in China
Brief Title: Clinical Investigation of Oral Malodor for Max Fresh Toothpaste Containing Zinc Citrate Versus a Commercially Available Regular Fluoride Toothpaste
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2026-02-OMO-MFX-YPZ
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Oral Malodor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 (Experimental): Subjects will brush their teeth for two (2) minutes each time, twice daily (morning and evening), using the assigned study toothpaste according to the manufacturer's instructions for three (3) weeks.
  Interventions: Drug: Max Fresh Toothpaste
- Control toothpaste (Active Comparator): Subjects will brush their teeth for two (2) minutes each time, twice daily (morning and evening), using the assigned study toothpaste according to the manufacturer's instructions for three (3) weeks.
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Max Fresh Toothpaste — 0.5% zinc citrate
  Arms: Test 1
Drug: Colgate Cavity Protection Toothpaste — sodium fluoride
  Arms: Control toothpaste

SUMMARY:
The objective of this three-week clinical research study is to evaluate oral malodor for a toothpaste containing zinc citrate as compared to a commercially available regular fluoride toothpaste using the organoleptic method.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years, inclusive.
* Availability for the full three-week duration of the study.
* Good general health.
* Initial mean oral malodor (organoleptic) score ≥ 6.0 and ≤ 8.4.
* Signed informed consent form.

Exclusion Criteria:

* Presence of orthodontic bands.
* Tumors of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (e.g., purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five (5) or more carious lesions requiring immediate restorative treatment.
* Use of antibiotics within one (1) month prior to study entry.
* Participation in any other clinical study or test panel within one (1) month prior to study entry.
* Dental prophylaxis within two (2) weeks prior to the initial examination.
* History of allergies to oral care/personal care products or their ingredients.
* Use of prescription medications that might interfere with study outcomes.
* Medical condition that prevents fasting (no food or drink) for up to four (4) hours.
* History of drug and/or alcohol abuse.
* Pregnant or lactating (self-reported).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
organoleptic method | baseline, 3 weeks
  assessed using the 1-9 organoleptic scale